CLINICAL TRIAL: NCT06523855
Title: Clinical and Radiographic Evaluation of Bilateral Alveolar Cleft Grafting With Micro Plate Stabilization Versus Conventional Grafting Technique: A Preliminary Clinical Trial
Brief Title: Evaluation of Bilateral Alveolar Cleft Grafting With Micro Plate Stabilization Versus Conventional Grafting Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Ahmed Ibrahim Ahmed, Resident at oral and maxillofacial surgery department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4623358
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Cleft
Keywords: alveolar cleft; iliac crest grafting; microplate; bone resorption; oronasal fistula
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral alveolar cleft grafting using iliac crest particulate and microplate fixation (Experimental): in bilateral alveolar cleft, the cancellous particulate bone graft from anterior iliac crest will be used to fill the defect, 8-hole microplates will be used to fix the premaxilla using screws.
  The microplates are to be removed 6 to 9 months postoperatively.
  Interventions: Procedure: bilateral alveolar cleft grafting using iliac crest particulate and microplate fixation
- bilateral alveolar cleft grafting using iliac crest particulate (Active Comparator): in bilateral alveolar cleft, the cancellous particulate bone graft from anterior iliac crest will be used to fill the defect.
  Interventions: Procedure: bilateral alveolar cleft grafting using iliac crest particulate and microplate fixation

INTERVENTIONS:
Procedure: bilateral alveolar cleft grafting using iliac crest particulate and microplate fixation — bilateral alveolar cleft grafting using particulate iliac crest graft accompanied with fixation of graft and premaxilla using microplate

SUMMARY:
The aim of the study is to enhance the maxillary segments stability during graft healing using microplate fixation to be compared with conventional grafting technique regarding gained bone quality and quantity.

DETAILED DESCRIPTION:
In conventional cleft grafting technique, there is always risk for grafted bone resorption and recurrence of fistula formation. So alveolar cleft grafting using anterior iliac crest bone particles combined with microplate fixation of maxillary segments will work more efficient and prevent the fore mentioned risk of graft resorption and recurrence of fistula.

In conventional cleft grafting techniques, most of the cases reported in literature raised a debate regarding the final gained amount of bone, with subsequent recurrence of oronasal fistula. In this study, alveolar cleft grafting using anterior iliac crest bone particles combined with microplate fixation of maxillary segments and the conventional grafting technique will be compared to evaluate which technique will offer better reconstruction of the alveolar ridge with maintained bone width and height.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral complete maxillary alveolar cleft at the age of mixed dentition (between 9 and 12 years old).
* repaired cleft lip.
* Patients with medical history that did not hinder surgical intervention and have adequate proper oral hygiene.
* Both genders males and females will be included.

Exclusion Criteria:

* General contraindications to surgical intervention of the area.
* Patients with unilateral maxillary alveolar cleft.
* Patients with ill repaired cleft lip that will hinder the appropriate reconstruction of the alveolar cleft
* Subjected to irradiation in the head and neck area less than 1 year before surgery.
* Untreated periodontitis.
* Poor oral hygiene.
* Uncontrolled diabetes.
* Immunosuppressed or immunocompromised.
* Active infection or severe inflammation in the area intended for graft placement
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Unable to attend a 9-month follow-up.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Bone density immediate versus 6 months postoperatively. | 6 months
  bone density changes are measured using CBCT after 6 months via HU

SECONDARY OUTCOMES:
Bone width and height immediate versus 6 months postoperatively | 6 months
  bone height and width changes are measured using CBCT after 6 months in mm

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Mekhemer, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smarius B, Loozen C, Manten W, Bekker M, Pistorius L, Breugem C. Accurate diagnosis of prenatal cleft lip/palate by understanding the embryology. World J Methodol. 2017 Sep 26;7(3):93-100. doi: 10.5662/wjm.v7.i3.93. eCollection 2017 Sep 26. PMID 29026689
- [Background] Seifeldin SA. Is alveolar cleft reconstruction still controversial? (Review of literature). Saudi Dent J. 2016 Jan;28(1):3-11. doi: 10.1016/j.sdentj.2015.01.006. Epub 2015 Jun 25. PMID 26792963
- [Background] Mahardawi B, Boonsiriseth K, Pairuchvej V, Wongsirichat N. Alveolar cleft bone grafting: factors affecting case prognosis. J Korean Assoc Oral Maxillofac Surg. 2020 Dec 31;46(6):409-416. doi: 10.5125/jkaoms.2020.46.6.409. PMID 33377466
- [Background] Boyne PJ, Sands NR. Secondary bone grafting of residual alveolar and palatal clefts. J Oral Surg. 1972 Feb;30(2):87-92. No abstract available. PMID 4550446
- [Background] Chen S, Liu B, Liu J, Yin N, Wang Y. Comparison of Three-Dimensional Printing and Computer-aided Engineering in Presurgical Volumetric Assessment of Bilateral Alveolar Clefts. J Craniofac Surg. 2020 Mar/Apr;31(2):412-415. doi: 10.1097/SCS.0000000000006011. PMID 31764559